CLINICAL TRIAL: NCT03132831
Title: Influence of the Operative Day on the Average Duration of Stay in Primary Hip and Knee Replacements
Acronym: JourOpDMS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: RNI2016-34 Pr Mertl
Record Dates: First submitted 2017-04-14; First posted 2017-04-28 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Length of Stay; Arthroplasty
MeSH Terms: interventions — Teniposide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Determine the DMS of the Total Hip Prosthesis of the University Hospital of Amiens (PTH) and the Total Knee Prosthesis (PTG) — To determine the DMS of the orthopedic department of the Amiens University Hospital after Total Hip Prosthesis (PTH) and First-line Total Knee Prosthesis (PTG) with its confidence interval and to compare it according to the patient's day of operation

SUMMARY:
Reducing the length of stay (LOS) after primary arthroplasty is a relatively new target that arouses the attention of orthopedic surgeons in order to return home early through the fast recovery protocols but this goal is also wanted in public health for the sake of overall decline health spending in public costs.

DETAILED DESCRIPTION:
Reducing the length of stay (LOS) after primary arthroplasty is a relatively new target that arouses the attention of orthopedic surgeons in order to return home early through the fast recovery protocols but this goal is also wanted in public health for the sake of overall decline health spending in public costs.

Reducing the LOS after primary hip arthroplasty and knee is studied through many publications that found an LOS influenced by the own medical factors of patients (ref) However, no study to our knowledge research the influence of the operative day and the LOS.

For historical reasons, the organization of care is modified on the weekend (Saturday and Sunday) in particular by reducing the caregiver and also the lack of physical therapist to make the early postoperative get up (D0 or D1).

The hypothesis is that a patient operated the friday did not have the same care the first 48 hours that a patient who had surgery at the beggening of the week and that his recovery was therefore extended.

The investigator can also suppose that LOS was shorter for patients returning home for those who were transferred to a rehabilitation center or other structure.

The results will be adjusted according to the literature data on the age more than 80 years, sex, diabetes, cardiovascular diseases, respiratory diseases.

ELIGIBILITY:
Inclusion Criteria:

* All major patients operated at the University Hospital of Amiens between 1 January 2015 and 31 December 2016 for primary hip and knee arthroplasty

Exclusion Criteria:

* All patients undergoing surgery for hip or knee surgery (reoperation).
* All patients undergoing total arthroplasty on fracture of the femoral neck from all causes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing primary hip and knee arthroplasty
Sampling Method: Non-Probability Sample
Enrollment: 1663 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Analysis of the average length of stay in total hip and knee arthroplasty (defined as the time in days between in and out of the orthopedic unit for all destinations) | 1 year
  Analysis of the average length of stay in total hip and knee arthroplasty (defined as the time in days between in and out of the orthopedic unit for all destinations)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France